CLINICAL TRIAL: NCT04154826
Title: Recombinant Interleukin-7 (CYT107) to Treat Patients With Refractory Nontuberculous Mycobacterial Lung Disease. Two Doses Phase II, Single Center, Open-label Trial
Brief Title: Recombinant Interleukin-7 (CYT107) to Treat Patients With Refractory Nontuberculous Mycobacterial Lung Disease
Acronym: IMPULSE-7
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: non convincing results
Sponsor: Revimmune (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPULSE-7
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — Interleukin-7

STUDY DESIGN:
Intervention Model Description: Two dose level parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose (Experimental): CYT107 10µg/kg/week for 4 weeks (wk1-4) followed by no treatment during 4 weeks (wk 5-8) CYT107 10µg/kg/week for 4 weeks (wk9-12)
  Interventions: Drug: Recombinant human interleukin-7
- high dose (Experimental): CYT107 20µg/kg/week for 4 weeks (wk1-4) followed by no treatment during 4 weeks (wk 5-8) CYT107 20µg/kg/week for 4 weeks (wk9-12)
  Interventions: Drug: Recombinant human interleukin-7

INTERVENTIONS:
Drug: Recombinant human interleukin-7 — weekly intra-muscular (IM) administration
  Other Names: CYT107

SUMMARY:
A prospective, single-center, single-blinded study involving patients with refractory nontuberculous mycobacteria lung disease to ascertain pharmacokinetics, safety, efficacy, and tolerability of two dose levels of parenteral administration of recombinant Interleukin-7 (IL-7) (CYT107).

DETAILED DESCRIPTION:
A single center, randomized, phase II, single blinded, two-dose level trial aimed at testing anti-mycobacterial activity of CYT107 in patients with non-tuberculous mycobacteria lung disease (NTMLD).

A total of 12 evaluable NTMLD patients from Washington University School of Medicine in St. Louis will be recruited and randomized 6:6 to study drug treatment at either 10μg/kg/wk or 20μg/kg/wk for two 4-week treatment periods.

The randomization will be stratified based on the presence of pulmonary cavitaries. A maximum of three patients with pulmonary cavitary disease will be allocated to each group.

A potential study extension is envisioned in the United Kingdom, in which case the protocol would be amended to increase the targeted enrollment and number of participating centers.

The aim of this trial is detection of an immuno-therapeutic response in patients with refractory NTMLD and to determine the potential rate of response and tolerance of CYT107 using two dose levels that indicated good immune response in other pathologies such as HIV, HCV, sepsis and various cancers.

For patients with refractory NTMLD, a control group is not beneficial as the standard of care treatment results are already known and documented.

All serious adverse events (SAEs) will be reported within 24 hours of notification

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years but <85 years who have given written informed consent to participate
2. Diagnosis of pulmonary nontuberculous mycobacterial lung disease in accordance with the 2007 Infectious DiseasesSociety of America (IDSA) and AmericanThoracic Society (ATS) criteria with evidence of nodular bronchiectatic and/or cavitary disease by chest CT
3. History of chronic, refractory infection with either Mycobacterium avium complex, defined as:

   1. Persistently positive mycobacterial sputum cultures after 6 or more months of guideline-based treatment (GBT), with at least one positive sputum culture within 2 months prior to the baseline visit and
   2. Currently on a stable guideline-based therapy that has been unchanged for the past 28 days. (GBT defined as a multi-drug regimen containing a macrolide and at least one other antimicrobial with activity against NTM.)
4. Ability to produce at least 3 mL of sputum or be willing to undergo an induction to produce at least 3 mL of sputum for clinical evaluation
5. This study permits the re-enrollment of a participant who may have been discontinued as a pre-treatment screen failure prior to study drug treatment.
6. Age and reproductive status:

   1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment
   2. Women must not be breastfeeding
   3. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with CYT107 plus 5 half-lives of CYT107 (the terminal half-life of CYT107 is up to 2 days) plus 30 days (duration of ovulatory cycle) for a total of 2 months post-treatment completion.
   4. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with CYT107 plus 5 half-lives of CYT107 plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
   5. Azoospermic males are exempt from contraceptive requirements.
   6. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements but still must undergo pregnancy testing as described in this section.

Exclusion Criteria:

1. Cancer with current chemotherapy or radiotherapy (receipt of chemotherapy or radiotherapy for cancer within the last 6 months). All patients with current, or history of, hematologic malignancy (including, but not limited to, acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), chronic lymphocytic leukemia (CLL), chronic myeloid leukemia (CML), etc.) or lymphoma will be excluded, regardless of receipt of recent chemotherapy
2. Active pulmonary tuberculosis requiring concomitant treatment at the time of screening
3. Patients with history or current evidence of autoimmune disease including for example: myasthenia gravis, Guillain Barre syndrome, systemic lupus erythematosus, multiple sclerosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's etc.
4. Patients who have received solid organ transplant or bone marrow transplant
5. Known history of infection with HIV or HIV positive test at screening
6. Known history of chronic HBV (hepatitis B viral) infection and not on treatment with HBV nucleoside analogues prior to the current hospitalization or HBV DNA > 100 IU/mL
7. Known history of infection with HCV (hepatitis C virus) and currently undergoing treatment for HCV infections or has detectable HCV RNA
8. History of splenectomy
9. Any hematologic disease associated with hypersplenism, such as thalassemia, hereditary spherocytosis, Gaucher's Disease, and autoimmune hemolytic anemia
10. Significant liver or renal dysfunction as evidence by at least 5 times greater than the upper limits of normal baseline ALT (alanine aminotransferase), AST (aspartate aminotransferase), alkaline phosphatase, or total bilirubin.
11. Evidence of biliary cirrhosis with portal hypertension
12. Participation in another investigational interventional study testing a drug or a medical device concurrently or within the last 28 days prior to study entry
13. Patients receiving immunosuppressive drugs or concurrent immunotherapy or biologic agents; including: growth factors, cytokines and interleukins other than the study medication: Interleukin-2, Interferons α, β and γ, GM-CSF, G-CSF (colony stimulating factors), HIV vaccines, biologics including TNF alpha inhibitors (i.e. abatacept, adalimumab, anakinra, certolizumab, etanercept, golimumab, infliximab, ixekizumab, natalizumab, rituximab, secukinumab, tocilizumab, ustekinumab, vedolizumab, basiliximab and daclizumab), calcineurin inhibitors, mammalian target of rapamycin inhibitors, inosine monophosphate dehydrogenase inhibitors, Janus kinase inhibitors, hydroxyurea, immunoglobulins, adoptive cell therapy
14. Patients receiving corticosteroids at a dose greater than 300mg hydrocortisone/ day or 25 mgs of prednisone per day or equivalent for more than 3 weeks
15. Prior exposure to exogenous IL 7
16. Inability to comply with the study treatment, study visits, and study procedures as assessed by the study PI or delegate
17. Subjects with hemoptysis of ≥60 mL in a 24 hour period within 4 weeks prior to screening
18. Addition of any new antimicrobial drug with known activity against Mycobacterium avium complex infection (i.e. amikacin, azithromycin, bedaquiline, clarithromycin, ciprofloxacin, clofazimine, ethambutol, eravacycline, levofloxacin, linezolid, moxifloxacin, omadacycline, rifampin, rifabutin, tedizolid, tigecycline tobramycin) within 28 days prior to Study Day 1
19. Daily continuous oxygen supplementation >4 L/min
20. Patients unlikely to survive a minimum of 30 days defined by (Systolic blood pressure) SBP<90 or hypoxia <80% SpO2 (oxygen saturation) -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Determination of the proportion of subjects with Acid Fast Bacilli (AFB) sputum culture conversion to negative at day 180. | six months
  Percentage of participants with 3 consecutive monthly, negative Acid Fast Bacilli sputum cultures at any time within first 6 months

SECONDARY OUTCOMES:
Efficacy by kinetic of AFB sputum culture conversion to negative. | one year
  number of patients with negative sputum conversion measured at days 28, 56, 84, 112, 140, 180, 240, 300, and 360.
Improvement of functional capacity response assessed by the median change in the 6-minute walk distance compared to baseline. | one year
  Increase in 6-minute walking distance measured at days 84, 180 and 360 over baseline distance
Improvement of functional capacity response assessed by the median change in oxygen saturation compared to baseline. | one year
  Increase in oxygen saturation measured at days 84, 180 and 360 over baseline value
Pulmonary function response measured by the median improvement in the Forced expiratory volume during the first second (FEV1). | one year
  ratio of Forced Expiratory Volume during the first second (FEV1) measured at days 180 and 360 over the same measure at baseline.
Radiological response on chest CT compared to baseline | one year
  Surface area of lung involved by clinical chest computerized tomography (CT) scans at days 180 and 360 compared to baseline
Improvement of Health-related Quality of Life (HRQoL) | one year
  Patient-Reported Outcomes Measurement Information System (PROMIS-29 ) measured at days 56, 84, 180, 300 and 360 and compared to baseline.
  (The mean healthy population score is 50. The score increases with worsening medical condition.)
Number of hospital readmissions | one year
  Cumulated Number of hospital (Intensive care unit or emergency room ) visits at days 56, 84, 180, 300 and 360
C max (maximal plasma concentration) pharmacokinetic of CYT107 in this population | One day
  At Day 1 and Day 78 measure of CYT107 Cmax
Plasma concentration area under curve (AUC) pharmacokinetic of CYT107 in this population | One day
  At Day 1 and Day 78 measure of CYT107 AUC
Clinical tolerance of CYT107 indicated by the study drop-out rate (%) regardless of the cause. | six months
  Percentage of patients who dropout of the study at days 28, 84, 180
Proportion of patients developing any grade 3-4 adverse events or deaths | one year
  Percentage of patients with grade 3-4 adverse events (assessed by CTCAE version 5.0) or deaths through day 360.
Measure of CYT107 immunogenicity | 1 year
  Number of patients with presence of binding and neutralizing antibodies at day 15, 29, 57, 90 and 120 compared to baseline. Testing for immunogenicity will be repeated at day 180 and again at day 360 only if positive antibodies are detected at previous sampling timepoint.

OTHER OUTCOMES:
IL-7 effect on opportunistic bacterial, viral or fungal infections | one year
  The incidence of new bacterial, fungal, or viral infections requiring medical treatment will be quantitated and captured during the interim history at each visit through Day 360.
IL-7 Effects on immune cells counts | one year
  The absolute lymphocyte, monocyte, and neutrophil counts will be assessed and compared to baseline values at days 28, 56, 84, 180 and one year (about day 360)
IL-7 Effects on CD4+ and CD8+ T lymphocytes | one year
  The absolute CD4+ and CD8+ T cell counts will be assessed and compared to baseline values at days 28, 56, 84, 180 and one year (about day 360)
IL-7 Effects on immune T cell markers | 2 months
  Peripheral blood cellular immune biomarkers including CD4 and CD8 T cell expression of soluble IL-7 receptor α (CD127), PD-1, and Ki67 and monocyte HLA-DR expression will be assessed at baseline and days 28, 56
IL-7 Effects on circulating cytokines | 2 months
  Circulating cytokines including Tumor necrosis factor (TNF-α), IL-6, and IL-10 will be measured by ELISA at baseline, Day 1 and day 56
IL-7 Effects on cellular cytokine production | 3 months
  ELISpot assays for stimulated production of Interferon (IFN-γ) and TNF-α will be performed at baseline and days 28, 56 and 84

CONTACTS AND LOCATIONS:
Overall Officials: Andrej SPEC, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mejia-Chew C, Spec A, Walton AH, Ulezko Antonova A, Dram A, Bhalla S, Colonna M, Morre M, Hotchkiss R. Recombinant interleukin-7 treatment of refractory Mycobacterium avium complex lung disease (IMPULSE-7): a pilot phase II, single-center, randomized, clinical trial. Ther Adv Infect Dis. 2025 May 10;12:20499361251339300. doi: 10.1177/20499361251339300. eCollection 2025 Jan-Dec. PMID 40351870